CLINICAL TRIAL: NCT02041000
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intravenously in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Adipose Derived Cells for Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Bioheart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-US-COPD-001
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pulmonary; stem cells; emphysema; lungs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

INTERVENTIONS:
Other: Adipose Derived Stem Cells

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* A prior diagnosis of moderate or severe COPD
* GOLD III and IV
* Age between 18 and 85 years

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. will have an expert consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Severe asthma that would contraindicate surgery
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Patients with Alpha-1
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 months
  Safety will be assessed as the occurrence/frequency (if applicable) of adverse events during the study procedures and for up to 6 months afterward.
St. George Respiratory | 6 months
  The St. George Respiratory questionnaire is an index developed to identify the quality of life of patients by measuring and quantifying health-related health status of patients with airflow obstruction.

SECONDARY OUTCOMES:
Gold Classification | 6 months
  The GOLD COPD staging system classifies people with COPD based on their degree of airflow limitation (obstruction). The airflow limitation is measured during pulmonary function tests
6 Minute Walk Test | 6 months
  Exercise capacity as measured as the distance a patient can walk over a 6 minute time period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Comella, Study Director — Bioheart
Locations (1):
- US Stem Cell Clinic, Sunrise, Florida, United States